CLINICAL TRIAL: NCT03418038
Title: Phase2 Trial of High Dose Intravenous Ascorbic Acid as an Adjunct to Salvage Chemotherapy in Relapsed/ Refractory Lymphoma, Patients With Clonal Cytopenia of Undetermined Significance, and Chronic Myelomonocytic Leukemia
Brief Title: Ascorbic Acid and Chemotherapy for the Treatment of Relapsed or Refractory Lymphoma, CCUS, and Chronic Myelomonocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LS1781; P50CA097274 (NIH); NCI-2018-00057 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LS1781 (Other: Mayo Clinic in Rochester); 17-008096 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Clonal Cytopenia of Undetermined Significance; High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Hodgkin Lymphoma; Recurrent Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Lymphoma; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Lymphoma; Leukemia, Myelomonocytic, Chronic | interventions — Ascorbic Acid; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Etoposide; Gemcitabine; Ifosfamide; Oxaliplatin; Rituximab; CT-P10; Decitabine; Injections; Specimen Handling; Biopsy, Needle; Biopsy, Large-Core Needle; Biopsy; Magnetic Resonance Spectroscopy; X-Rays; Central Venous Catheters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (ascorbic acid, combination chemotherapy) (Experimental): Patients receive ascorbic acid IV on days 1, 3, 5, 8, 10, 12, 15, 17, and 19, and rituximab intravenously IV, ifosfamide IV, carboplatin IV and etoposide IV on days 1-3. Patients who achieve MR or SD after 2 cycles may receive rituximab IV or PO, cisplatin IV or PO, cytarabine IV or PO, and dexamethasone IV or PO. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients additionally, undergo blood sample collection, core needle biopsy, bone marrow aspiration and biopsy, ECHO, PET/CT or MRI throughout study.
  Interventions: Dietary Supplement: Ascorbic Acid; Drug: Carboplatin; Drug: Cisplatin; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Biological: Rituximab; Procedure: Biospecimen Collection; Procedure: Core Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography
- Arm B (placebo, combination chemotherapy) (Active Comparator): Patients receive placebo (normal saline) IV on days 1, 3, 5, 8, 10, 12, 15, 17, and 19, and rituximab intravenously IV, ifosfamide IV, carboplatin IV and etoposide IV on days 1-3. Patients who achieve MR or SD after 2 cycles may receive rituximab IV or PO, cisplatin IV or PO, cytarabine IV or PO, and dexamethasone IV or PO. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients additionally, undergo blood sample collection, core needle biopsy, bone marrow aspiration and biopsy, ECHO, PET/CT or MRI throughout study.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Questionnaire Administration; Biological: Rituximab; Procedure: Biospecimen Collection; Procedure: Core Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography
- Arm C (ascorbic acid and combination chemotherapy) (Experimental): Patients receive ascorbic acid IV on days 1, 3, 5, 8, 10, 12, 15, 17, and 19. Patients also receive ifosfamide, carboplatin, and etoposide IV or PO, or cisplatin, cytarabine, and dexamethasone IV or PO, or gemcitabine hydrochloride, dexamethasone, and cisplatin IV or PO, or gemcitabine hydrochloride and oxaliplatin IV or PO, or oxaliplatin, cytarabine, and dexamethasone IV or PO according to standard regimen schedule. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve MR or SD after 2 cycles may switch to an alternative chemotherapy regimen. Patients additionally, undergo blood sample collection, core needle biopsy, bone marrow aspiration and biopsy, ECHO, PET/CT or MRI throughout study.
  Interventions: Dietary Supplement: Ascorbic Acid; Drug: Carboplatin; Drug: Cisplatin; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Gemcitabine Hydrochloride; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Oxaliplatin; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Procedure: Core Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography
- Arm D (ascorbic acid) (Experimental): Patients receive ascorbic acid IV TIW. Treatments repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo PICC or portacath placement prior to starting treatment, blood sample collection, bone marrow aspiration and biopsy throughout study.
  Interventions: Dietary Supplement: Ascorbic Acid; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Central Venous Cannula Insertion; Procedure: Portacath Placement
- ARM E (ascorbic acid, decitabine) (Experimental): Patients receive ascorbic acid IV on days 1, 3 and 5 and decitabine IV over 1 hour on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 12 cycles may continue decitabine with or without ascorbic acid as long as clinically appropriate. Patients may also take vitamin C PO on days 6-28. Patients undergo PICC or portacath placement prior to starting treatment, blood sample collection, bone marrow aspiration and biopsy throughout study.
  Interventions: Dietary Supplement: Ascorbic Acid; Drug: Decitabine; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Central Venous Cannula Insertion; Procedure: Portacath Placement

INTERVENTIONS:
Dietary Supplement: Ascorbic Acid — Given IV
  Other Names: 2-(1,2-dihydroxyethyl)-4,5-dihydroxy-furan-3-one; Asorbicap; C Vitamin; C-Long; Ce-Vi-Sol; Cecon; Cenolate; Cetane; Cevalin; L-Ascorbic Acid; VIT C; Vitamin C; Vitamin-C
  Arms: ARM E (ascorbic acid, decitabine); Arm A (ascorbic acid, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy); Arm D (ascorbic acid)
Drug: Carboplatin — Given IV or PO
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo; JM8
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Drug: Cisplatin — Given IV or PO
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Drug: Cytarabine — Given IV or PO
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Drug: Etoposide — Given IV or PO
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16-213; VP16; VP-16
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Drug: Gemcitabine Hydrochloride — Given IV or PO
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY-188011; LY188011
  Arms: Arm C (ascorbic acid and combination chemotherapy)
Drug: Ifosfamide — Given IV or PO
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy); Arm D (ascorbic acid)
Drug: Oxaliplatin — Given IV or PO
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
  Arms: Arm C (ascorbic acid and combination chemotherapy)
Other: Placebo Administration — Given normal saline IV
  Arms: Arm B (placebo, combination chemotherapy)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy); Arm D (ascorbic acid)
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Riabni; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-pvvr; RTXM83; Ruxience; Truxima; Ikgdar; Mabtas
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy)
Drug: Decitabine — Given IV
  Other Names: Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
  Arms: ARM E (ascorbic acid, decitabine)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Core Biopsy — Undergo core needle biopsy
  Other Names: BIOPSY, CORE; CORE CNB; Core Needle; Core Needle Biopsy; Needle Biopsy
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC; ECHO
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; nuclear magnetic resonance imaging; Structural MRI; sMRI
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)
Procedure: Central Venous Cannula Insertion — Undergo PICC placement
  Other Names: Central venous catheter; Central Venous Catheter Placement
  Arms: ARM E (ascorbic acid, decitabine); Arm D (ascorbic acid)
Procedure: Portacath Placement — Undergo portacath placement
  Other Names: Port-a-cath Placement
  Arms: ARM E (ascorbic acid, decitabine); Arm D (ascorbic acid)
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT SCAN; tomography
  Arms: Arm A (ascorbic acid, combination chemotherapy); Arm B (placebo, combination chemotherapy); Arm C (ascorbic acid and combination chemotherapy)

SUMMARY:
This phase II trial studies the effect of ascorbic acid and combination chemotherapy in treating patients with lymphoma that has come back (recurrent) or does not respond to therapy (refractory), clonal cytopenia of undetermined significance and chronic myelomonocytic leukemia (CMML). Ascorbic acid may make cancer cells more sensitive to chemotherapy. Drugs used in chemotherapy, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ascorbic acid and combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate (ORR) at the end of 2 cycles for intravenous (IV) ascorbic acid (AA) added to standard salvage therapy compared to standard salvage therapy plus normal saline in patients with relapsed/refractory diffuse large B-cell lymphoma (DLBCL) who have relapsed within the first 24 months of end of their therapy. [Arms A versus (vs) B] II. To determine the ORR at the end of 2 cycles of AA plus standard salvage chemotherapy in patients with other types of relapsed/refractory lymphomas not eligible for Arms A/B [peripheral T-cell lymphoma (PTCL), double-hit high grade, and Hodgkin lymphoma (HL)]. (Arm C) III. To assess the hematological response rate to treatment with high dose intravenous ascorbic acid (IV AA) for clonal cytopenia of undetermined significance (CCUS) patients. (Arm D) IV. To assess the hematological response rate to treatment with high dose intravenous ascorbic acid (IV AA) for CCUS patients. (Arm E)

SECONDARY OBJECTIVES:

I. To compare the adverse event profile of IV AA added to salvage therapy versus salvage therapy plus IV saline in patients with DLBCL using both the Common Terminology Criteria for Adverse Events (CTCAE) and Patient-Reported Outcomes (PRO)-CTCAE. (Arms A and B) II. To compare the progression-free survival, overall survival, clinical benefit rate (those not progressing), and percentage (%) transplant eligible patients proceeding to transplant of AA added to salvage therapy versus salvage therapy plus IV saline in patients with DLBCL. (Arms A and B) III. To compare the ORR at the end of 4 cycles for those with minor response/stable disease at the end of cycle 2 who proceed to receive the additional 2 cycles of rituximab, dexamethasone, cytarabine and cisplatin (RDHAP) with either AA or normal saline (NS) as previously assigned. (Arms A and B) IV. To evaluate the adverse event profile, rate of febrile neutropenia, overall survival, progression-free survival, and clinical benefit rate of AA added to salvage therapy in patients with relapsed/refractory lymphoma. (Arm C) V. To assess safety/tolerability, transfusion dependency (TD), progression-free survival (PFS), and overall survival (OS) for CCUS patients receiving high dose IV AA. (Arm D) VI. To define CR, complete cytogenetic remission, partial remission, marrow response, and clinical benefit response rates. (Arm E) VII. To determine clinical benefit response rates of erythroid response, platelet response, neutrophil response, spleen response and symptom response as adjudicated by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) total symptom scoring system. (Arm E)

EXPLORATORY OBJECTIVES:

I. Will include baseline AA levels [at Mayo Clinic Research (MCR)] and staining of pre/post treatment biopsies for markers of oxidative stress generation and deoxyribonucleic acid (DNA) methylation. (Arms A, B, and C Correlative Research on blood and tumor tissue) IIa. To assess TET2 activity at baseline, weeks 12, 20, and 52. (Arm D correlative research) IIb. To assess the association between using AA and the hydroxymethylation and methylation status (gene-specific and global changes in 5mC/5hmC level) at baseline and weeks 20 and 52. (Arm D correlative research) IIc. To assess the association between using IV AA and endothelial dysfunction (at baseline, weeks 20, and 52). (Arm D correlative research) IId. To assess the association between using IV AA and the inflammation markers. (Arm D correlative research) IIe. To assess the association between using IV AA and molecular response including clonal dynamics [new mutations and variant allele frequency (VAF)] (at baseline, weeks 20, and 52). (Arm D correlative research)

III. Correlative studies will assess impact on:

IIIa. Somatic mutational allele burdens after 4 cycles of therapy; IIIb. DNA methylation and hydroxymethylation after 4 cycles of therapy; IIIc. Inflammatory cytokines; IIId. Colony forming assay growth and differentiation; IIIe. Methylation at the single colony level; IIIf. Single cell methylation, transcription, and somatic mutations. (Arm E correlative research)

OUTLINE: Patients with DLBCL are randomized to Arms A or B. Patients with other lymphomas are assigned to Arm C. Patients with CCUS are assigned to Arm D. Patients with TET2 mutant CMML are assigned to ARM E.

Arm A: Patients receive ascorbic acid IV on days 1, 3, 5, 8, 10, 12, 15, 17, and 19, and rituximab intravenously (IV), ifosfamide IV, carboplatin IV and etoposide IV on days 1-3. Patients who achieve minor response (MR) or stable disease (SD) after 2 cycles may receive rituximab IV or PO, cisplatin IV or PO, cytarabine IV or PO, and dexamethasone IV or PO. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive placebo (normal saline) IV on days 1, 3, 5, 8, 10, 12, 15, 17, and 19, and rituximab intravenously IV, ifosfamide IV, carboplatin IV and etoposide IV on days 1-3. Patients who achieve MR or SD after 2 cycles may receive rituximab IV or PO, cisplatin IV or PO, cytarabine IV or PO, and dexamethasone IV or PO. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive ascorbic acid IV on days 1, 3, 5, 8, 10, 12, 15, 17, and 19. Patients also receive ifosfamide, carboplatin, and etoposide IV or PO, or cisplatin, cytarabine, and dexamethasone IV or PO, or gemcitabine hydrochloride, dexamethasone, and cisplatin IV or PO, or gemcitabine hydrochloride and oxaliplatin IV or PO, or oxaliplatin, cytarabine, and dexamethasone IV or PO according to standard regimen schedule. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve MR or SD after 2 cycles may switch to an alternative chemotherapy regimen.

ARM D: Patients receive ascorbic acid IV three times a week (TIW). Treatments repeat every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

ARM E: Patients receive ascorbic acid IV on days 1, 3 and 5 and decitabine IV over 1 hour on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease after 12 cycles may continue decitabine with or without ascorbic acid as long as clinically appropriate. Patients may also take vitamin C PO on days 6-28.

In Arms A, B, and C, patients who achieve complete response (CR), partial response (PR) or MR may undergo stem cell transplantation. Patients additionally, undergo blood sample collection, core needle biopsy, bone marrow aspiration and biopsy, echocardiography (ECHO), positron emission tomography (PET)/ computed tomography (CT) or magnetic resonance imaging (MRI) throughout study.

Patients in ARM D and E undergo peripherally inserted central catheter (PICC) or portacath placement prior to starting treatment, blood sample collection, bone marrow aspiration and biopsy throughout study.

After completion of study treatment, patients are followed up every 3 months, then every 6 months after progressive disease for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Biopsy-proven relapsed or refractory lymphomas; relapsed is defined as a relapse that occurred after having a response to the last therapy that lasted > 6 months; refractory is no response or relapse within 6 months; previous biopsies < 6 months prior to treatment on this protocol will be acceptable

  * NOTE: Arms A/B - relapsed or refractory DLBCL within 24 months from the end of anthracycline-based therapy; no prior salvage therapy; patients can have received radiation therapy as part of initial treatment but not specifically for relapse
  * NOTE: Arm C patients include relapsed or refractory lymphoma patients of any type for which the recommended treatment includes one of the platinum-based regimens; of note, relapsed or refractory double-hit high grade lymphoma patients and relapsed or refractory Hodgkin lymphoma patients will be enrolled in Arm C; there is no limit on the number of prior therapies for Arm C patients; the patient must be eligible for a platinum-based regimen and must not have received the same regimen in the past without responding
* Measurable or assessable disease: measurable disease is defined as measurable by computed tomography (CT) [dedicated CT or the CT portion of a positron emission tomography (PET)/CT] or magnetic resonance imaging (MRI): to be considered measurable, there must be at least one lesion that has a single diameter of >= 1.5 cm

  * NOTE: Skin lesions can be used if the area is >= 1.5 cm in at least one diameter and photographed with a ruler; patients with assessable disease by PET are also eligible as long as the assessable disease is biopsy proven lymphoma
* Arms A/B - eligible for treatment with ifosfamide, carboplatin, and etoposide (+/- rituximab)
* Arm C eligible for treatment with one of the following standard, every 3 week, platinum-based salvage regimens (with or without monoclonal antibody as appropriate for the disease):

  * Ifosfamide/carboplatin/etoposide (ICE) or rituximab/ifosfamide/carboplatin/etoposide (RICE);
  * Cisplatin, cytarabine (cytosine arabinoside), dexamethasone (DHAP) or RDHAP;
  * Gemcitabine hydrochloride (gemcitabine), dexamethasone, cisplatin (GDP) or rituximab, gemcitabine, dexamethasone, cisplatin (RGDP);
  * Gemcitabine and oxaliplatin (GemOx) or rituximab, gemcitabine and oxaliplatin (RGemOx);
  * Oxaliplatin, cytosine arabinoside, dexamethasone (OAD) or rituximab, oxaliplatin, cytosine arabinoside, dexamethasone (ROAD)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Hemoglobin >= 8.0 g/dL (may transfuse to meet this requirement), obtained =< 14 days prior to registration
* Absolute neutrophil count (ANC) >= 1500/mm^3, obtained =< 14 days prior to registration
* Platelet count >= 75000/mm^3, obtained =< 14 days prior to registration
* Total bilirubin =< 2 x upper limit of normal (ULN) (if > 2 x ULN direct bilirubin is required and should be =< 1.5 x ULN), obtained =< 14 days prior to registration
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement), obtained =< 14 days prior to registration
* Creatinine =< 1.6 mg/dL; if over 1.6 then the calculated creatinine clearance must be >= 55 ml/min using the Cockcroft-Gault formula, obtained =< 7 days prior to registration
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Human immunodeficiency virus (HIV) test done =< 14 days prior to registration

  * If positive, the CD4 count must be > 400
* Provide written informed consent
* Willingness to have a central venous line [peripherally inserted central catheter (PICC) or PORT]
* Willingness to provide mandatory blood specimens for correlative research
* Willingness to provide mandatory tissue specimens for correlative research
* Willingness to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willingness to follow the requirements of the intravenous ascorbic acid program schedule
* ARM D: Patients who had a diagnosis of CCUS with one or more TET2 mutations or TET2 mutations with concurrent splicing genes mutations (SRSF2, U2AF1, SF3B1, and ZRSR2) or epigenetic regulator mutations (DNMT3A, EZH2, IDH1, IDH2). CCUS diagnosis being defined based on the absence of definitive morphologic evidence of hematologic neoplasms from bone marrow biopsy evaluation combined with evidence of pathogenic myeloid somatic mutation with a variant allele frequency (VAF) of at least 2% using our institution's next generation sequencing (NGS) panel (OncoHeme, Mayo Clinic)
* ARM D: ECOG performance status (PS) 0, 1 or 2
* ARM D: Patients must meet at least 1 of these 3 laboratory criteria to be enrolled:

  * Hemoglobin =< 10g/dL (obtained =< 7 days prior to registration)
  * Absolute neutrophil count (ANC) =< 1000/mm^3 (obtained =< 7 days prior to registration)
  * Platelet count =< 100,000/mm^ 3 (obtained =< 7 days prior to registration)
* ARM D: Total bilirubin =< 2 x ULN (if > 2 x ULN direct bilirubin is required and should be =< 1.5 x ULN) (obtained =<7 days prior to registration)
* ARM D: Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 3 x ULN (=< 5 x ULN for patients with liver involvement) (obtained =<7 days prior to registration)
* ARM D: Creatinine =< 1.6 mg/dL (obtained =<7 days prior to registration). If > 1.6, then the Calculated creatinine clearance must be >= 55 ml/min using the Cockcroft-Gault formula
* ARM D: Negative pregnancy test, for persons of childbearing potential only (obtained =< 7 days prior to registration). NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* ARM D: Provide written informed consent
* ARM D: Willingness to have a central venous line (PICC or PORT)
* ARM D: Willingness to provide mandatory blood specimens for correlative research
* ARM D: Willingness to return to enrolling institution (MCR) for follow-up (during the active monitoring phase of the study)
* ARM D: Willingness to follow the requirements of the intravenous ascorbic acid program schedule
* ARM E PRE-REGISTRATION: Age ≥ 18 years
* ARM E PRE-REGISTRATION: New or an established diagnosis of 2016 World Health Organization (WHO) defined chronic myelomonocytic leukemia with a somatic TET2, IDH1, or IDH2 mutation requiring treatment with DNA methyltransferase inhibitors/hypomethylating agents
* ARM E PRE-REGISTRATION: No prior CMML directed therapy.

  * Exception: Received ≤ 1 cycle of azacitidine, decitabine, erythropoiesis stimulating agent therapy (ESA), or oral decitabine and cedazuridine. NOTE: Prior exposure to hydroxyurea is allowed. Continuation beyond the first cycle must be discussed with the principal investigator (PI)
* ARM E PRE-REGISTRATION: Creatinine ≤ 1.6 mg/dL. If > 1.6, then the Calculated creatinine clearance must be ≥ 55 ml/min using the Cockcroft-Gault formula
* ARM E PRE-REGISTRATION: Willingness to provide mandatory research bone marrow sample for correlative research
* ARM E PRE-REGISTRATION: ECOG performance status (PS) 0, 1, or 2
* ARM E PRE-REGISTRATION: Provide written informed consent
* ARM E REGISTRATION: Willingness to provide mandatory blood specimens for correlative research
* ARM E REGISTRATION: Willingness to return to enrolling institution (MCR) for follow-up (during the active monitoring phase of the study)
* ARM E REGISTRATION: Recovered to grade 1 or baseline or established as sequelae from all toxic effects of previous therapy except alopecia
* ARM E REGISTRATION: Absolute neutrophil count (ANC) ≥ 500/mm^3 (obtained ≤ 7 days prior to registration)
* ARM E REGISTRATION: Platelet count ≥ 20,000/mm^3 (obtained ≤ 7 days prior to registration)
* ARM E REGISTRATION: Total bilirubin ≤ 1.5 x ULN ( ≤ 3 x ULN for patients with Gilbert's syndrome) (obtained ≤ 7 days prior to registration)
* ARM E REGISTRATION: Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (obtained ≤ 7 days prior to registration)
* ARM E REGISTRATION: Ability to complete questionnaire by themselves or with assistance
* ARM E REGISTRATION: For a person of child-bearing potential (WOCBP): Must agree to use contraception or take measures to avoid pregnancy during the study. Adequate contraception is defined as follows:

  * Complete true abstinence
  * Consistent and correct use of one of the following methods of birth control:

    * Male partner who is sterile prior to the female patient's entry into the study and is the sole sexual partner for that female patient
    * Implants of levonorgestrel
    * Injectable progestogen
    * Intrauterine device (IUD) with a documented failure rate of less than 1% per year
    * Oral contraceptive pill (either combined or progesterone only)
    * Barrier method, for example: diaphragm with spermicide or condom with spermicide in combination with either implants of levonorgestrel or injectable progestogen
* ARM E REGISTRATION: WOCBP must have a negative serum or urine pregnancy test ≤ 7 days prior to registration. NOTE: WOCBP include any person who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea > 12 consecutive months); or women on hormone replacement therapy with documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL. Even women who are using oral, implanted, or injectable contraceptive hormones or mechanical products such as an IUD or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy or practicing abstinence or where partner is sterile (e.g., vasectomy), must be considered to be of child-bearing potential. NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* ARM E REGISTRATION: Persons who are able to father a child must use contraception during the study and for 3 months after the last treatment dose.

  * Complete true abstinence
  * Latex condom with a spermicidal agent
  * Diaphragm with spermicide
* ARM E REGISTRATION: Willingness to have a central venous line (PICC or PORT)
* ARM E REGISTRATION: Willingness to follow the requirements of the intravenous ascorbic acid program schedule

Exclusion Criteria:

* Any of the following:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Any therapy =< 2 weeks prior to registration; NOTE: Exception: patients on ibrutinib or corticosteroids (any dose) may continue therapy up until the new regimen has started at investigator discretion; corticosteroids can be tapered to lowest possible dose after start of treatment at investigator discretion. Exception: Palliative radiation is allowed
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, pulmonary congestion or pulmonary edema, clinical dehydration, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the lymphoma
* Other active malignancy than lymphoma

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer that could interfere with this protocol therapy; patients on hormonal therapy for treated breast or prostate cancer are permitted if they meet other eligibility criteria; patients with non-melanotic skin cancer may enroll
* History of myocardial infarction =< 6 months, or current symptomatic congestive heart failure or left ventricular ejection fraction (LVEF) < 40% or with > grade 2 diastolic dysfunction, with no symptoms or signs of heart failure
* Known G6PD (glucose-6-phosphate dehydrogenase) deficiency (below lower limit of normal)
* Patients with active central nervous system (CNS) lymphoma or active cerebrospinal fluid (CSF) involvement with malignant cells requiring CNS-specific therapy with IV or intrathecal (IT) methotrexate (MTX); Note: Patients with any prior CNS lymphoma (parenchymal or leptomeningeal) MUST be in complete remission (CR) in those compartments without any maintenance therapy required
* Patients with uncontrolled or symptomatic kidney stones
* Known paroxysmal nocturnal hemoglobinuria (PNH)
* ARM D: Bona-fide hematological neoplasm
* ARM D: Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* ARM D: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* ARM D: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, pulmonary congestion or pulmonary edema, clinical dehydration, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* ARM D: History of myocardial infarction =< 6 months, or current symptomatic congestive heart failure or known LVEF < 40% or with > grade 2 diastolic dysfunction, with no symptoms or signs of heart failure
* ARM D: Patients with uncontrolled or symptomatic kidney stones
* ARM D: Known paroxysmal nocturnal hemoglobinuria (PNH)
* ARM D: Known G6PD (glucose-6-phosphate dehydrogenase) deficiency (below lower limit of normal)
* ARM E PRE-REGISTRATION: Myelodysplastic syndrome (MDS)/myeloproliferative neoplasm (MPN) overlap syndromes other than CMML
* ARM E PRE-REGISTRATION: Active central nervous system disease
* ARM E PRE-REGISTRATION: Any active disease condition that would render the protocol treatment dangerous or impair the ability of the patient to receive study drug
* ARM E PRE-REGISTRATION: Concurrent active malignancy, except adequately treated nonmelanoma skin cancer. History of curatively treated in situ cancer of the cervix, curatively treated in situ cancer of the breast, or other solid tumors curatively treated is allowed as long as there is no evidence of disease for > 2 years
* ARM E PRE-REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* ARM E PRE-REGISTRATION: Disease requiring systemic treatment with systemic immunosuppression with steroid steroids at a dose of ≥ 20 mg/day prednisone (or equivalent). Exceptions: Intermittent use of bronchodilators or inhaled steroids, local steroid injections, topical steroids
* ARM E PRE-REGISTRATION: Patients with uncontrolled or symptomatic kidney stones
* ARM E REGISTRATION: New York Heart Association (NYHA) class III/IV heart failure or active angina/angina equivalents
* ARM E REGISTRATION: History of myocardial infarction ≤ 6 months, or current symptomatic congestive heart failure or known LVEF < 40% or with > grade 2 diastolic dysfunction, with no symptoms or signs of heart failure
* ARM E REGISTRATION: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant cardiac arrhythmia, unstable angina pectoris, clinically significant nonhealing or healing wounds, pulmonary congestion or pulmonary edema, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection, clinical dehydration, or psychiatric illness/social situations that would limit compliance with study requirements
* ARM E REGISTRATION: Known G6PD (glucose-6-phosphate dehydrogenase) deficiency (below lower limit of normal)
* ARM E REGISTRATION: Any of the following because this study involves an agent that has known genotoxic, mutagenic, and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (Arms A and B) | Up to 2 years
  Defined as an objective status of complete response (CR) or partial response (PR) evaluated by Response Evaluation Criteria in Lymphoma (RECIL) criteria after 2 courses of treatment in all arms. Will be compared between the two arms. The proportion of successes will be estimated in each arm by the number of successes divided by the total number of evaluable patients. Exact binomial ninety-five percent confidence intervals for the true success proportion will be calculated in each arm. For the diffuse large B-cell lymphoma (DLBCL) arms, comparison of overall response rates between the two treatment groups will be performed using a one-sided chi-square test at significance level 0.10.
ORR (Arm C) | Up to 2 years
  Defined as an objective status of CR or PR evaluated by RECIL criteria after 2 cycles of treatment. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Exact binomial ninety-five percent confidence intervals for the true success proportion will be calculated in each arm.
Hematologic response (HI) rate (Arm D) | At 20 weeks
  Defined as an objective status of HI-E (minor or major response), HI-P, or HI-N evaluated by Myelodysplastic Syndrome International Working Group (IWIG) 2018 criteria at 20 weeks. Exact binomial ninety-five percent confidence intervals for the true success proportion will be calculated in each arm.
Overall Response Rate (ORR) in Arm E | At completion of cycle 4 (each cycle is 21 days)
  Defined as an objective status of complete remission, complete cytogenetic remission, partial remission, bone marrow response, or clinical benefit after 4 cycles of therapy as defined by the 2015 IWG myelodysplastic syndrome/ myeloproliferative neoplasm response criteria.

SECONDARY OUTCOMES:
Clinical benefit rate (Arms A, B, and C) | Up to 2 years
  Will be estimated in each arm by the number of patients who achieve a CR, PR, minor response (MR), or stable disease (SD) on the cycle 2 response assessment divided by the total number of evaluable patients. Exact binomial 95% confidence intervals for the true success rate will be calculated. The clinical benefit rate will be compared between the DLBCL arms using the chi-square test (or Fisher's exact test if the data in the contingency table is sparse).
Overall survival | From registration to death due to any cause, assessed up to 2 years
  The distribution of overall survival will be estimated in each arm using the method of Kaplan-Meier. In the DLBCL arms, the comparison of overall survival between the two treatment arms will be based on the log-rank test.
Progression-free survival | From date of first treatment to the earliest date of documentation of disease progression or death due to any cause, assessed up to 2 years
  The distribution of progression-free survival will be estimated in each arm using the method of Kaplan-Meier. In the DLBCL arms, the comparison of progression-free survival between the two treatment arms will be based on the log-rank test.
Percent of transplant eligible patients proceeding to transplant (Arms A, B and C) | Up to 2 years
  Will be estimated in each arm by the number of patients proceeding to transplant divided by the total number of patients who were considered transplant eligible. Exact binomial 95% confidence intervals for the true success rate will be calculated. The rate will be compared between the DLBCL arms using the chi-square test (or Fisher's exact test if the data in the contingency table is sparse).
Transfusion dependency (Arm D) | Up to 2 years
  Transfusion dependency will be summarized descriptively. The number of patients transfusion dependent at baseline and during follow-up will be summarized.
Incidence of adverse events | Up to 2 years
  Assessed using Common Terminology Criteria for Adverse Events (CTCAE). The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. In the DLBCL arms, the overall adverse event rates for Grade 3 or higher hematologic and non-hematologic adverse events at least possibly related to treatment will be compared between the two treatment groups using the chi-square test (or Fisher's exact test if the data in the contingency table is sparse). The rate of febrile neutropenia will be evaluated in each arm.
Incidence of adverse events | Up to 2 years
  Assessed using Patient Reported Outcomes (PRO)-CTCAE (Arms A and B). PRO-CTCAE scores range from 0-4, with corresponding response choices for frequency (Never / Rarely / Occasionally / Frequently / Almost constantly), for severity (None / Mild / Moderate / Severe / Very severe) and interference (Not at all / A little bit / Somewhat / Quite a bit / Very much). The scores for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. PRO-CTCAE scores will be compared between the two treatment groups using the chi-square test (or Fisher's exact test if the data in the contingency table is sparse).
Continued salvage therapy beyond cycle 2 (Arm A, B and C) | Up to 2 years
  Will be assessed by evaluating the number of patients who achieve an improved response after cycle 4 compared to the cycle 2 assessment in patients who received additional cycles of ascorbic acid/placebo added to salvage therapy beyond cycle 2. In addition, the number of patients who changed salvage therapies after cycle 2 will be assessed. This analysis will be primarily descriptive.
Clinical benefit rate (Arm E) | Up to 2 years
  The rates of complete response, complete cytogenetic remission, partial remission, marrow response, and clinical benefit will be estimated by the number of patients with each response type divided by the number of evaluable patients.
Hematologic response rate in Arm E | Up to 2 years
  The rates of erythroid response, platelet response, neutrophil response, spleen response and symptom response will be estimated by the number of patients with each response type divided by the number of evaluable patients.

OTHER OUTCOMES:
Biomarker analysis on blood and tissue (Arms A, B, and C) | Baseline up to 2 years
  Will consider the correlative research exploratory.
Biomarker analysis (Arm D) | Baseline up to 2 years
  Variant allele frequency (VAF), biomarkers levels from Olink study, values of the cytokines, endothelial dysfunction, inflammation markers and levels of 5mc/5hmc will be measured at baseline, after completion of treatment (at 20 weeks), and at one-year post-registration. Values will be summarized graphically and descriptively at each time point and changes across time will be explored. Due to small sample size, these correlative analyses will be considered exploratory.
Molecular response (Arm D) | Up to 2 years
  Defined as a 2 standard deviation reduction in VAF from baseline VAF. Exact binomial 95% confidence intervals for the true success rate will be calculated.
TET2 activity (Arm D) | At baseline and weeks 12, 20, 52
  Values will be summarized graphically and descriptively at each time point and changes across time will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Witzig, M.D., Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- [Derived] Xie Z, Fernandez J, Lasho T, Finke C, Amundson M, McCullough KB, LaPlant BR, Mangaonkar AA, Gangat N, Reichard KK, Elliott M, Witzig TE, Patnaik MM. High-dose IV ascorbic acid therapy for patients with CCUS with TET2 mutations. Blood. 2024 Dec 5;144(23):2456-2461. doi: 10.1182/blood.2024024962. PMID 39352751
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials